CLINICAL TRIAL: NCT05413785
Title: Prospective Cohort Study to Determine Effectiveness of Telemedicine-based on Site Hepatitis C Management in Probation and Parole Office
Brief Title: Hepatitis C Treatment in Probation and Parole Office
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rosenau (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Jens Rosenau, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IMDDN-22-HEP-C-TX
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-09

CONDITIONS: Hepatitis C; HCV
Keywords: parole; probation; telemedicine
MeSH Terms: conditions — Hepatitis C | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with Hepatitis C (Experimental): Participants will be clients at the Lexington Probation and Parole office who are Hepatitic C positive.
  Interventions: Behavioral: Telehealth in Parole/Probation Office

INTERVENTIONS:
Behavioral: Telehealth in Parole/Probation Office — Onsite (telehealth) linkage toHep C treatment in a Probation and Parole office setting via an onsite nurse navigator. The navigator will provide Hep C education, draw labs, and facilitate a telemed visit with a UK GI provider.

SUMMARY:
This prospective cohort study compares aims to determine the efficacy and effectiveness of telemedicine-supported on-site linkage to care and treatment in a community probation and parole office (P&P office) setting and compare the results with a historic control with referral to care. Research participants will be followed in the P&P office when they report to their officer during regularly scheduled appointments. Participants will receive treatment without having to travel to a specialist's office. The telemedicine visit will include a consultation with an experienced HCV provider such as a hepatologist or an advanced practice provider and a specialty pharmacist who will educate about and monitor HCV treatment. The UK specialty pharmacy will be available to participants and the HCV management team through a 24-hour support line. Participants will be treated per HCV guidelines and insurance preference.

ELIGIBILITY:
Inclusion Criteria:

* Clients who will be supervised in the probation and parole office for at least 5 months
* History of hepatitis C
* Able to obtain health insurance
* Capacity to provide written, informed consent
* Life expectancy >1 year

Exclusion Criteria:

* Negative HCV RNA
* Pregnant or breast-feeding
* HIV or HBV co-infection
* Liver cirrhosis with Child-Turcotte-Pugh score 6 or greater at baseline lab work
* Subjects with impaired capacity to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
HCV treatment uptake rate of HCV RNA positive participants | 6 months
  Percentage of treatment uptake among treatment eligible patients seen by a provider via telemedicine.

SECONDARY OUTCOMES:
HCV treatment uptake rate | 6 months
  percentage of all chronically infected patients regardless of treatment eligibility
Determine visit adherence | 6 months
  Number of kept visits divided by number of scheduled visits

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rosenau, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No